CLINICAL TRIAL: NCT05108987
Title: Exercise Time of Day for Cardiometabolic Health in Type 2 Diabetes
Brief Title: Exercise and Time of Day in Type 2 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Noom Inc. (Industry)
Responsible Party: Principal Investigator, Steven K Malin, PhD, Associate Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro2021001183
Record Dates: First submitted 2021-10-26; First posted 2021-11-05 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Diabetes Mellitus, Type 2; Metabolic Syndrome
Keywords: type 2 diabetes; diet; exercise; mobile application; cardiometabolic; metabolic health; behavioral; vascular health; blood flow; continuous glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Metabolic Syndrome; Motor Activity; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Morning Exercise (Experimental): If subjects are randomly assigned to this group, they will participate in exercise training in the morning at a moderate to hard intensity. Subjects will be asked to regularly engage in morning exercise while supervised for about 2 weeks.
  Interventions: Behavioral: Morning Exercise
- Afternoon Exercise (Active Comparator): If subjects are assigned to this group, they will participate in the same exercise program but after in the afternoon.
  Interventions: Behavioral: Afternoon Exercise

INTERVENTIONS:
Behavioral: Morning Exercise — Exercise at moderate to hard intensity will be performed in the morning for up to 10 sessions for about 1 hour under supervision in the morning.
  Arms: Morning Exercise
Behavioral: Afternoon Exercise — Exercise at moderate to hard intensity will be performed in the morning for up to 10 sessions for about 1 hour under supervision in the afternoon.
  Arms: Afternoon Exercise

SUMMARY:
The overall purpose of the study is to test the effect of Noom on exercise and diet advice in adults with type 2 diabetes. The overarching hypothesis is that the use of Noom may promote better dietary adherence during an exercise program, thereby promoting greater weight loss and cardiometabolic health compared to lifestyle advice only. In particular, the investigators anticipate that changes in metabolic and vascular insulin sensitivity will correlate with glycemic control and blood pressure changes.

DETAILED DESCRIPTION:
Type 2 diabetes (T2D) is associated with a 3-fold cardiovascular disease (CVD) mortality risk compared with healthy controls, and it is estimated that 30 million adults in the United States have the disease. In recent years the American Diabetes Association (ADA) and American College of Sports Medicine (ACSM) recommend moderate intensity (40-60% heart rate max, HRmax) aerobic exercise 3-5d/wk for the management of T2D. The statement also recognized that higher exercise intensity (>60% HRmax) predicts better blood glucose control than exercise volume. Cardiovascular health (e.g. fitness, blood pressure, etc.) also appears to respond in an exercise dose dependent manner. Despite these suggestions, many people exercising compensate by eating calories back from exercise, thereby negating weight loss. Moreover, compliance and adherence to exercise and diet medical counsel is disappointingly low.

Recent work has begun to target the best time of day to exercise in effort to improve weight loss and related health. This has evolved in part since circadian biology reveals people tend to become glucose intolerant, and develop insulin resistance and endothelial dysfunction in the evening compared with morning. As a result, it would be reasonable to hypothesize that exercise in the afternoon may be best at combating natural declines in health as well as optimizing training adaptations. However, not all studies agree that afternoon is the best time to exercise. In fact, some have demonstrated that 12 wks of aerobic plus resistance exercise improved glycemic control whether performed in the morning or afternoon in adults with T2D. Moreover, consistent morning exercise has been suggested to improve exercise adherence through possible enjoyment as well as lead to greater weight loss. Taken together, additional work is warranted to understand time of day in which exercise is performed given circadian influence may contribute to variations in favorable metabolic as well as vascular adaptation for CVD prevention/treatment. Excitingly, we have preliminary data showing that afternoon exercise induces greater weight loss, reductions in food intake as well as perceptions of appetite and increased insulin sensitivity when compared to morning exercisers. Thus, the overall purpose of this proposal is to determine whether exercise time of day differentially enhances likelihood of weight loss via appetite regulation as well as glycemic control. Our overarching hypothesis is that afternoon exercise will enhance the effectiveness of exercise to induce weight loss, improve appetite and improve glycemic regulation compared to exercise in the morning. Taken together, findings from this study will inform public health recommendations to contemporary behavioral strategies to treat T2D. The study will also provide much needed experimental evidence to time of day in which exercise is performed influences public health risk.

ELIGIBILITY:
Inclusion Criteria:

* Male or female >30 and <70 years old.
* Has a body mass index >28 and <45 kg/m2.
* Previously diagnosed with T2DM.
* Subjects currently taking medications that affect heart rate and rhythm (i.e. Ca++ channel blockers, nitrates, alpha- or beta-blockers).

Exclusion Criteria:

* Morbidly obese patients (BMI >46 kg/m2) and overweight/lean patients (BMI <27 kg/m2)
* Evidence of type 1 diabetes and diabetics requiring insulin therapy
* Subjects who have not been weight stable (>2 kg weight change in past 3 months)
* Subjects who have been recently active (>30 min of moderate/high intensity exercise, 2 times/week).
* Subjects who are smokers or who have quit smoking <1 years ago
* Subjects with abnormal estimated glomerular filtration rate (eGFR).
* Hypertriglyceridemic (>400 mg/dl) and hypercholesterolemic (>260 mg/dl) subjects
* Hypertensive (>160/100 mmHg)
* Subjects with a history of significant metabolic, cardiac, congestive heart failure, cerebrovascular, hematological, pulmonary, gastrointestinal, liver, renal, or endocrine disease or cancer that in the investigator's opinion would interfere with or alter the outcome measures or impact subject safety.
* Pregnant (as evidenced by positive urine pregnancy test) or nursing women
* Subjects with contraindications to participation in an exercise training program
* Currently taking active weight suppression medication (e.g. phentermine,orlistat, lorcaserin, naltrexone-bupropion in combination, liraglutide, benzphetamine, diethylpropion, phendimetrazine)
* Known hypersensitivity to perflutren (contained in Definity)

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-09-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Body Weight | Over the course of 2 weeks.
  The primary outcome is changes in body weight pre- and post-intervention

SECONDARY OUTCOMES:
Glucose Tolerance | Over the course of 2 weeks.
  We will examine the influence of Noom on the glucose area under the curve during the oral glucose tolerance test.
Flow-mediated dilation | Over the course of 2 weeks.
  We will assess blood flow to better understand nutrient/glucose delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Steven K Malin, PhD, Principal Investigator — Rutgers University - New Brunswick
Locations (3):
- United States (3):
  - New Jersey Institute for Food, Nutrition, and Health, New Brunswick, New Jersey
  - Robert Wood Johnson University Hospital Clinical Research Center, New Brunswick, New Jersey
  - Rutgers University Loree Gymnasium, New Brunswick, New Jersey

IPD SHARING:
Plan to Share IPD: No